CLINICAL TRIAL: NCT00270465
Title: VRC101: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Prime-Boost HIV-1 Vaccination Schedule of a 6-Plasmid Multiclade HIV-1 DNA Vaccine, VRC-HIVDNA016-00-VP, Followed by a Recombinant Multiclade Adenoviral Vector HIV Vaccine
Brief Title: Safety and Immune Response to a Prime-Boost Vaccination Schedule in HIV-infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060056; 06-I-0056; NCT00255853 (obsolete NCT alias)
Record Dates: First submitted 2005-12-24; First posted 2005-12-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-06-25

CONDITIONS: HIV
Keywords: HIV-positive; Treatment Interruption; Therapeutic Vaccine; HIV/AIDS; Virologic Response; HIV Positive
MeSH Terms: conditions — HIV Seropositivity; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: VRC-HIVDNA016-00-VP
Drug: VRC-HIVADV014-00-VP

SUMMARY:
Study Design: This is a Phase I, randomized, placebo-controlled, double-blinded study to examine safety, tolerability and immune response of a prime-boost vaccination regimen for treatment of HIV infection. The vaccination schedule consists of three injections of a multiclade HIV plasmid DNA vaccine followed by one injection of a multiclade recombinant adenoviral vector vaccine (rAd), in HIV-infected adults. The hypothesis is that this vaccination regimen will be safe and elicit an immune response in HIV-infected subjects. The primary objectives are related to evaluating the safety and tolerability of the vaccination regimen and assessing the effect of vaccination on humoral and cellular immune responses to vaccine-specific HIV antigens.

Product Description: VRC-HIVDNA016-00-VP is composed of 6 closed, circular DNA plasmids that are each 16.67% (by weight) of the vaccine. Each of the 6 plasmids in this vaccine expresses a single gene product. Plasmids VRC 4401, VRC 4409 and VRC 4404 are designed to express clade B HIV-1 Gag, Pol and Nef, respectively. VRC 5736, VRC 5737, and VRC 5738 are designed to express HIV-1 Env glycoprotein from clade A, clade B, and clade C, respectively. Each DNA vaccination will be 1 mL of vaccine administered intramuscularly (IM) using the Biojector 2000 Needle-Free Injection Management System. Phosphate buffered saline (PBS) will be used as the placebo for the DNA vaccine.

VRC-HIVADV014-00-VP (rAd) is a recombinant product composed of 4 adenoviral vectors (Ad) (in a 3:1:1:1 ratio) that encode the HIV-1 Gag/Pol polyprotein from clade B and HIV-1 Env glycoproteins from clades A, B, and C, respectively. Injections of 10(10) PU will be administered IM by needle and syringe. The final formulation buffer (FFB) will be used as the placebo for the rAd vaccine.

Subjects: HIV-infected adult volunteers (18-50 years old) on stable highly active antiretroviral therapy (HAART) therapy who have a CD4+ cell count greater than 350 cells/mm3 and have had a viral load (VL) less than 400 copies/mL for at least six months and a viral load of less than 50 copies/mL within 4 weeks prior to enrollment.

Study Plan: Fifteen volunteers will be enrolled and randomized in a 2:1 ratio to vaccine:control (10 DNA prime with rAd boost:5 PBS with FFB placebo). A Data and Safety Monitoring Board (DSMB) will review the study every 6 months. Subjects will be evaluated for safety and immunogenicity for 48 weeks, which is 24 weeks after the target date for the booster vaccination.

Study Duration: Subjects will be followed for 48 weeks after enrollment into the study.

DETAILED DESCRIPTION:
This study will determine the safety and side effects of two experimental HIV vaccines and see if vaccination can enhance the pre-existing HIV-specific immune response in HIV-infected individuals on anti-retroviral therapy . The vaccines are VRC-HIVDNA016-00-VP (called the "DNA vaccine") and VRC-HIVADV014-00-VP (called the "rAd vaccine"). The DNA vaccine codes for four HIV proteins. The rAd vaccine is made using an adenovirus (a common virus that causes upper respiratory infections, such as the common cold) that has been modified to contain DNA that codes for three HIV proteins. These vaccines will be given in a "prime-boost" schedule and cannot cause HIV or adenoviral infections.

HIV-infected people between 18 and 50 years old who are on a stable treatment plan for HIV with highly active antiretroviral (ARV) drugs, have a CD4+ T cell count greater than 350, and have a low viral load may be eligible for this 48-week study.

Participants receive an injection (shot) of the DNA vaccine or a placebo (solution that does not contain any vaccine, medicine, or drugs) the day they enter the study and again at study weeks 4 and 8. They receive a booster injection of the rAd vaccine or placebo at week 24. The DNA vaccines are given with a needle-less injection device called the "Biojector 2000(Registered Trademark)" and the rAd vaccine is given using a needle and syringe. All shots are given in the upper arm muscle, alternating right and left arms with each injection. Patients fill out a diary card at home for 5 days after each vaccination, recording their temperature and any symptoms. The cards are turned in to the clinic at the first visit after all 5 days are completed. Patients must call a study nurse 1 or 2 days after each of the four injections and again 7 or 8 days after each of the first three injections.

Patients have 12 clinic visits during the course of the study. At each visit, they are checked for health changes or problems, asked how they are feeling and if they have taken any medications or other treatments, including over-the-counter medicines, herbal supplements, etc. Blood samples are drawn at every visit and urine samples are collected at some visits.

At week 28 (4 weeks after the fourth injection), patients undergo apheresis, a procedure for collecting large numbers of white blood cells. The cells are tested in the laboratory to see how the immune system responds to the study vaccine. For the procedures, blood is collected through a needle in an arm vein and spun in a machine that separates the white blood cells from the rest of the blood (red cells, plasma and platelets). The white cells are removed and the rest of the blood is returned to the patient's body through the same needle. Patients who cannot or do not want to undergo apheresis have 80 mL (about 1/3 cup) of blood drawn through a needle and collected in blood collection tubes.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. HIV-1 infection defined as documented by any approved ELISA test kit and confirmed with a Western blot at any time prior to study entry.
2. On stable highly active antiretroviral therapy (HAART), as defined by the Department of Health and Human Services (http://www.aidsinfo.nih.gov/other/cbrochure/english/04_en.pdf), with no change in the drugs included in the treatment regimen for a minimum of 8 weeks prior to enrollment.
3. CD4+ cell count greater than 350 cells/mm(3) at 2 different time points that meet the following criteria: The first result must be from between 4 weeks to 36 weeks prior to enrollment obtained at any laboratory used by a health care facility. The second result must be obtained at the NIH Clinical Center within 28 days prior to enrollment. There must be at least 28 days between the two tests used for eligibility.
4. HIV-1 RNA viral load (VL) consistently less than 400 copies/mL for six months or longer prior to enrollment (as reported by the subject). Documentation must include the following: at least one documented HIV RNA PCR result showing VL less than 400 copies/mL obtained between 12-36 weeks prior to enrollment at any laboratory used by a health care facility and another VL less than 50 copies/mL that must be obtained at the NIH Clinical Center within 28 days prior to study entry.
5. Men and women aged 18-50 years.
6. Ability and willingness of subject to give written informed consent.

   Laboratory Criteria within 28 days prior to enrollment:
7. Absolute neutrophil count (ANC) greater than or equal to 750/mm(3).
8. Hemoglobin greater than or equal to 9.0 g/dL.
9. Platelet count greater than or equal to 100,000/mm(3).
10. Creatinine less than or equal to 1.5 x upper limit of normal (ULN).
11. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x ULN.
12. Total bilirubin less than or equal to 2.5 x ULN; a higher total bilirubin value may be permitted if the subject is taking atanazir (ATV) or indinavir (IDV) and the elevation in total bilirubin is due to increased indirect (unconjugated) bilirubin.
13. Serum lipase less than or equal to 2.0 x ULN.
14. Normal urinalysis, defined as negative glucose, negative or trace protein, and no clinically significant blood in the urine.

    Female-Specific Criteria:
15. Female study volunteers of reproductive potential must have a negative serum or urine pregnancy test on the day of enrollment into the study. All female study participants are presumed to be of reproductive potential unless they have been post-menopausal for at least 24 consecutive months or have undergone surgical sterilization (e.g. hysterectomy, bilateral oophorectomy, or salpingotomy). If participating in sexual activity that could lead to pregnancy, the female study volunteer must use a form of contraception listed below starting at least 21 days prior to enrollment and continuing to Week 48 of the study. At least one of the following methods MUST be used appropriately (with or without hormone-based method):

Condoms (male or female) with or without a spermicidal agent;

Diaphragm or cervical cap with spermicide;

IUD.

If the female volunteer is not of reproductive potential as defined above she is eligible without requiring the use of contraception. Patient-reported history is acceptable as documentation of sterilization, contraceptive methods, or menopause.

EXCLUSION CRITERIA:

Women:

1. Breast-feeding or planning to become pregnant during the 48 weeks of study participation.

   A volunteer will be excluded if he/she has a medication history of one or more of the following:
2. Receipt of live attenuated vaccines or investigational research agents within 30 days prior to study entry.
3. Receipt of blood products within 120 days prior to study entry.
4. Receipt of immunoglobulin within 60 days prior to study entry.
5. Receipt of medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal, or allergy treatment with antigen injections) within 14 days prior to study entry.
6. Receipt of experimental HIV vaccines in the preceding 2 years. Individuals that received a placebo in a prior HIV vaccine trial are not excluded.
7. Receipt of immunosuppressive medications within the past 6 months (e.g., oral/parenteral/inhaled corticosteroids, and/or cytotoxic medications). NOTE: The following will be allowed: corticosteroid nasal spray for allergic rhinitis; topical corticosteroids for acute, uncomplicated dermatitis; over the counter medications for acute, uncomplicated dermatitis for a period not longer than 14 days; short-acting beta-agonists in controlled asthmatics; or a short course (10 days or less) of corticosteroids for a non-chronic condition at least 2 weeks prior to enrollment in the study.
8. Receipt of IL-2 within the preceding 1 year.

   A volunteer with any of the following conditions will be excluded:
9. Positive hepatitis B virus (HBV) surface antigen or positive hepatitis C virus (HCV) antibody or detectable HCV viral load.
10. History of CD4+ counts less than 100 cells/mm(3) on two or more occasions in the past.
11. History of serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. Subjects who have a history of an adverse reaction to pertussis vaccine as a child may enroll.
12. History of autoimmune disease; immunodeficiency (other than HIV infection); asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the prior 2 years or that requires the use of oral or intravenous corticosteroids; diabetes (Type I or II with the exception of gestational diabetes); thyroidectomy or history of thyroid disease in the past 12 months; or serious angioedema episodes within the previous 3 years or requiring medication in the previous 2 years.
13. Current antituberculosis-prophylaxis or therapy.
14. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
15. Serious illness (requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 14 days prior to study entry.
16. Hypertension that is not well controlled by medication or is more than 150/100 at enrollment.
17. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with intramuscular (IM) injections or blood draws.
18. Syphilis infection that is active or a positive serology due to a syphilis infection that has not been effectively treated.
19. Treated malignancy for which there is not reasonable assurance of sustained cure, or malignancy that required either lymph node irradiation or axillary dissection.
20. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.
21. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
22. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicide plan or attempt occurring within five years prior to enrollment.
23. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17
Dates: Start 2005-12-21; Primary Completion 2009-06-25 (Actual); Study Completion 2009-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Calmy A, Pascual F, Ford N. HIV drug resistance. N Engl J Med. 2004 Jun 24;350(26):2720-1. doi: 10.1056/NEJM200406243502621. No abstract available. PMID 15215494
- [Background] Clough LA, D'Agata E, Raffanti S, Haas DW. Factors that predict incomplete virological response to protease inhibitor-based antiretroviral therapy. Clin Infect Dis. 1999 Jul;29(1):75-81; discussion 82-4. doi: 10.1086/520185. PMID 10433568
- [Background] Lucas GM, Chaisson RE, Moore RD. Highly active antiretroviral therapy in a large urban clinic: risk factors for virologic failure and adverse drug reactions. Ann Intern Med. 1999 Jul 20;131(2):81-7. doi: 10.7326/0003-4819-131-2-199907200-00002. PMID 10419445
- [Derived] Casazza JP, Bowman KA, Adzaku S, Smith EC, Enama ME, Bailer RT, Price DA, Gostick E, Gordon IJ, Ambrozak DR, Nason MC, Roederer M, Andrews CA, Maldarelli FM, Wiegand A, Kearney MF, Persaud D, Ziemniak C, Gottardo R, Ledgerwood JE, Graham BS, Koup RA; VRC 101 Study Team. Therapeutic vaccination expands and improves the function of the HIV-specific memory T-cell repertoire. J Infect Dis. 2013 Jun 15;207(12):1829-40. doi: 10.1093/infdis/jit098. Epub 2013 Mar 12. PMID 23482645